CLINICAL TRIAL: NCT06908096
Title: Phase 1 Study of the Safety of an Epstein-Barr Virus (EBV) gH/gL/gp42-Ferritin Nanoparticle Vaccine With or Without gp350-Ferritin in Healthy Adults With or Without EBV Infection
Brief Title: Epstein-Barr Virus (EBV) gH/gL/gp42-Ferritin Nanoparticle Vaccine With or Without gp350-Ferritin in Healthy Adults With or Without EBV Infection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10002288; 002288-I
Record Dates: First submitted 2025-04-02; First posted 2025-04-03 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09-23

CONDITIONS: EBV; Epstein-Barr Virus Infection; Infectious Mononucleosis; Mono
Keywords: Infectious Mononucleosis; Neutralizing Antibody; Vaccine; EBV; Mono; Immune Response
MeSH Terms: conditions — Epstein-Barr Virus Infections; Infectious Mononucleosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental): There will be an initial dose escalation phase comprised of 9 EBV seropositive individuals.
  Interventions: Biological: EBV gp350-ferritin vaccine with ALFQ adjuvant; Biological: EBV gH/gL/gp42-ferritin nanoparticle vaccine with ALFQ adjuvant
- Randomization (Experimental): In the randomization phase, twenty-four EBV-seropositive individuals will be randomized in a 1:1 ratio to receive either 3 doses of adjuvanted gH/gL/gp42-ferritin alone or adjuvanted gH/gL/gp42-ferritin + gp350-ferritin nanoparticle.
  Interventions: Biological: EBV gp350-ferritin vaccine with ALFQ adjuvant; Biological: EBV gH/gL/gp42-ferritin nanoparticle vaccine with ALFQ adjuvant

INTERVENTIONS:
Biological: EBV gp350-ferritin vaccine with ALFQ adjuvant — The adjuvanted gH/gL/gp42-ferritin nanoparticle vaccine is given with gp350-ferritin intramuscularly into the deltoid muscle at 0, 1, and 4 months.
Biological: EBV gH/gL/gp42-ferritin nanoparticle vaccine with ALFQ adjuvant — The adjuvanted gH/gL/gp42-ferritin nanoparticle vaccine is given with gp350-ferritin intramuscularly into the deltoid muscle at 0, 1, and 4 months.

SUMMARY:
Background:

Epstein-Barr virus (EBV) is the primary cause of infectious mononucleosis, commonly known as mono. EBV infects more than 90% of the world s population. Mono can be serious, and it can lead to severe illnesses like cancer and autoimmune diseases. Researchers want to test vaccines that may help prevent EBV and associated diseases.

Objective:

To test two EBV vaccines: EBV gH/gL/gp42-ferritin and EBV gp350-ferritin.

Eligibility:

Healthy EBV-negative or EBV-positive people aged 18 to 29.

Design:

Participants will be screened. They will have a physical examination. They will give blood and saliva samples.

They will receive 3 doses of the study vaccine as an injection in the shoulder muscle. They will get either one vaccine or a combination of both vaccines.

Participants will get their first dose of the vaccine at visit 1, the second dose about 30 days later, and the final dose about 90 days after that.

Participants will be given a memory aid so they can record any symptoms and side effects between visits. This can be done either on paper or online through a link that is emailed to them.

There are 6 required in-person visits. There are also 2 optional visits. In between the in-person visits are 7 telehealth visits or phone calls. Each visit may take up to 4 hours.

The study will last for about 17 months. Participants will have the option of staying in the study for an additional year.

DETAILED DESCRIPTION:
Study Description:

This is a phase 1 study to evaluate the safety of a 3-dose vaccination regimen of an adjuvanted EBV gH/gL/gp42-ferritin nanoparticle vaccine with or without gp350-ferritin. Based on data reported in animal studies, our hypothesis is that this EBV vaccine will induce a potent immune response that neutralizes EBV infection of B cells and epithelial cells.

There will be an initial dose escalation phase comprised of 9 EBV-seropositive individuals followed by a randomization phase comprised of 24 EBV-seropositive individuals and an additional 30 EBV-seronegative individuals. In each group, the vaccine will be given at 0, 1, and 4 months, and participants will be followed until at least 12 months after the third dose of vaccine with an option to be followed for an additional year. Some individuals will receive only the EBV gH/gL/gp42-ferritin nanoparticle vaccine; others will receive EBV gH/gL/gp42-ferritin nanoparticle vaccine plus the gp350-ferritin nanoparticle vaccine. Participants will know which vaccine they have received during the study.

Objectives:

Primary objective: To determine the safety of an adjuvanted EBV gH/gL/gp42-ferritin nanoparticle vaccine with or without gp350-ferritin nanoparticle in seronegative and seropositive healthy adults.

Key secondary objective: To evaluate the immunogenicity of an adjuvanted EBV gH/gL/gp42-ferritin nanoparticle vaccine with or without gp350-ferritin nanoparticle in seronegative and seropositive healthy adults.

Endpoints:

Primary endpoints:

* Local and systemic vaccine side effects during the 7-day period after each vaccination
* All symptoms and diagnoses up to 30 days after each vaccination
* Serious medical events (SAEs) through 30 days after the last dose of study vaccine.

Key secondary endpoints:

-Production of EBV neutralizing antibody after the vaccination series, as measured by B cell and epithelial cell neutralization assays.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. 18 to 29 years old.
2. Able to provide informed consent.
3. Willingness to allow storage of blood and saliva for future research.
4. In good general health as evidenced by medical history, physical examination, and laboratory screening results.
5. Participant is willing to forgo receipt of a licensed, live vaccine in the 30 days preceding each dose of vaccine or in the 30 days following each dose of vaccine. Any FDA-approved inactivated, subunit, or replication-defective vaccine (such as COVID-19, influenza, tetanus, etc.) can be used >=14 days before or >=14 days after administration of the study vaccine.
6. Participants of reproductive potential who are sexually active with a partner who can impregnate them: use of highly effective continuous contraception for at least 30 days prior to Day 0 and agreement to continue use until 60 days after the last dose of vaccine.

Contraceptive requirements: Because the effects of EBV gH/gL/gp42-FNP and EBV gp350-ferritin vaccines on the developing human fetus are unknown, sexually active participants of childbearing potential must agree to use highly effective contraception as outlined below before study entry and until 60 days after the last dose of vaccine. Participants of childbearing potential must have a negative pregnancy test before receiving each dose of the EBV gH/gL/gp42-FNP vaccine. During the course of the study, if a participant becomes pregnant or suspects they are pregnant, then they should inform the study staff and their primary care physician immediately.

Acceptable forms of contraception are:

* Intrauterine device (IUD) or equivalent.
* Hormonal contraceptive (eg, consistent, timely, and continuous use of contraceptive pill, patch, ring, implant, or injection that has reached full efficacy prior to dosing). If the participant uses a contraceptive pill, patch, or ring, then a barrier method (eg, internal/external condom, cap, or diaphragm plus spermicide) must also be used at the time of potentially reproductive sexual activity.
* A stable, long-term monogamous relationship with a partner who does not pose any potential pregnancy risk, eg, has undergone a vasectomy at least 6 months prior to the first dose of vaccine or is of the same sex as the participant.
* A hysterectomy and/or a bilateral tubal ligation or bilateral oophorectomy.

Acceptable forms of contraception for participants who can impregnate a partner include one of the following:

* External condom plus spermicide, used during sexual intercourse, even if the partner uses a contraceptive pill, patch, or ring.
* A vasectomy completed at least 6 months before the first dose of vaccine.
* Continuously and completely abstaining from sexual intercourse with a partner of childbearing potential from the first dose of vaccine until 30 days after the last dose.

Acceptable contraception for partners of childbearing potential of participants who can impregnate them include one of the following:

* IUD or equivalent.
* Hormonal contraceptive (eg, pill, patch, ring, implant, or an injection used consistently and that has reached full effect prior to the first dose of vaccine).
* Hysterectomy and/or a bilateral tubal ligation or bilateral oophorectomy.

Laboratory Criteria within 30 days or less prior to enrollment:

1. Hemoglobin within institutional normal limits or if not, then assessed and deemed not clinically significant by PI or designee
2. White blood cell count and differential either within institutional normal reference range or if not then assessed and deemed not clinically significant by PI or designee
3. Total lymphocyte count (lymphocyte absolute) > 800 cells/microL
4. Platelet count equal to 125,000-500,000/microL
5. Alanine aminotransferase <1.25 x upper limit of normal (ULN)
6. Serum IgG >600 mg/dL

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pregnant, breastfeeding, or planning to become pregnant while participating through 60 days after the last dose of vaccine.
2. Participant has received any of the following:

   1. More than 10 days of systemic immunosuppressive medications (>=10 mg prednisone dose or its equivalent) or cytotoxic medication within the 30 days prior to first dose of vaccine or immunomodulating therapy within 180 days prior to first dose of vaccine.
   2. Blood products, including immunoglobulin products, within 120 days prior to first dose of vaccine.
   3. Investigational research agents within 30 days prior to first dose or planning to receive investigational products while on study.
   4. Allergy treatment with antigen injections, unless on a maintenance schedule of shots no more frequently than once per month.
   5. Prior participant in an EBV vaccine clinical trial.
3. Participant has any of the following:

   1. Febrile illness within 14 days of the first dose of vaccine.
   2. Body habitus such that it is difficult to confirm location of the deltoid muscle for safe intramuscular injection.
   3. History of serious reactions to vaccines.
   4. Hereditary, acquired, or idiopathic forms of angioedema.
   5. Idiopathic urticaria within the past year.
   6. Asthma that is not well-controlled or required emergent care, urgent care, hospitalization, or intubation during the past 2 years or that requires the use of oral or intravenous steroids.
   7. Diabetes mellitus type 1 or type 2, excluding a history of gestational diabetes.
   8. Clinically significant autoimmune disease or immunodeficiency.
   9. Hypertension that is not well-controlled.
   10. Thyroid disease that is not well-controlled.
   11. Bleeding disorder diagnosed by doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions).
   12. Significant bruising or bleeding difficulties with intramuscular injections or blood draws.
   13. Malignancy that is active or treated malignancy for which there is no reasonable assurance of sustained cure or malignancy that is likely to recur during the study period.
   14. Seizure disorder other than a history of 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the past 3 years.
   15. Asplenia, functional asplenia, or any condition resulting in absence or removal of the spleen.
   16. History of Guillain-Barre Syndrome.
   17. Alcohol or drug abuse or addiction.
   18. HIV infection.
4. Any medical, psychiatric, or social condition that, in the judgement of the investigator, is a contraindication to protocol participation or impairs the participant's ability to give informed consent.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Local and systemic reactogenicity signs and symptoms during the 7-day period after each vaccination. Unsolicited AEs up to 30 days after each vaccination and SAEs through Day 150. | Through Day 150
  To determine the safety of an adjuvanted EBV gH/gL/gp42-ferritin nanoparticle vaccine with or without gp350-ferritin nanoparticle in seronegative and seropositive healthy adults.

SECONDARY OUTCOMES:
Change in log10 antibody response to EBV from baseline to 30 days after the last dose of vaccine (Day 150) as measured by the B cell neutralization assay. | Through Day 150
  To evaluate the immunogenicity of an adjuvanted EBV gH/gL/gp42-ferritin nanoparticle vaccine with or without gp350 ferritin nanoparticle in seronegative and seropositive healthy adults.
Change in log10 antibody response to EBV from baseline to 30 days after the last dose of vaccine (Day 150) as measured by the epithelial cell neutralization assay. | Through Day 150
  To further evaluate the immunogenicity of the adjuvanted EBV gH/gL/gp42-ferritin nanoparticle vaccine with or without gp350-ferritin.
ELISA-determined dilution for for antibodies to H. pylori and/or human ferritin on Day 0, Day 30, Day 60, and Day 150. | Length of the study
  To determine whether the vaccine causes production of antibodies to H. pylori and/or human ferritin.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica R Durkee-Shock, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We allow sharing of essentially all de-identified data per the data sharing plan.
Supporting Information: ICF, CSR
Time Frame: Data will be shared after conclusion of the trial and upon request by appropriate researchers.
Access Criteria: Data will be shared in compliance with the NIH data sharing policy, the clinical protocol, and participant consent forms. Furthermore, sharing of data must also be approved by WRAIR.

REFERENCES:
- [Background] Cohen JI. Epstein-barr virus vaccines. Clin Transl Immunology. 2015 Jan 23;4(1):e32. doi: 10.1038/cti.2014.27. eCollection 2015 Jan. PMID 25671130
- [Background] Kanekiyo M, Bu W, Joyce MG, Meng G, Whittle JR, Baxa U, Yamamoto T, Narpala S, Todd JP, Rao SS, McDermott AB, Koup RA, Rossmann MG, Mascola JR, Graham BS, Cohen JI, Nabel GJ. Rational Design of an Epstein-Barr Virus Vaccine Targeting the Receptor-Binding Site. Cell. 2015 Aug 27;162(5):1090-100. doi: 10.1016/j.cell.2015.07.043. Epub 2015 Aug 13. PMID 26279189
- [Background] Wei CJ, Bu W, Nguyen LA, Batchelor JD, Kim J, Pittaluga S, Fuller JR, Nguyen H, Chou TH, Cohen JI, Nabel GJ. A bivalent Epstein-Barr virus vaccine induces neutralizing antibodies that block infection and confer immunity in humanized mice. Sci Transl Med. 2022 May 4;14(643):eabf3685. doi: 10.1126/scitranslmed.abf3685. Epub 2022 May 4. PMID 35507671
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002288-I.html